CLINICAL TRIAL: NCT00258037
Title: Six Months Follow-Up of Pelvic Floor Muscle Training in Women With Urinary Incontinence After Stroke
Brief Title: Effect of Pelvic Floor Muscle Training in Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST-KA98117
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2000-03

CONDITIONS: Stroke; Urinary Incontinence
Keywords: Physiotherapy; Stroke; Urinary Incontinence; quality of Life
MeSH Terms: conditions — Stroke; Urinary Incontinence

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle training

SUMMARY:
Aim: To evaluate the long term effect of pelvic floor muscle training in women with urinary incontinence after ischemic stroke measured by quality of life paramters.

ELIGIBILITY:
Inclusion Criteria:

* Female stroke patients
* one month since stroke
* UI in close relation to the stroke
* normal cognitive level
* independent walking indoor ability > 100 m
* independence in toilet visit

Exclusion Criteria:

* urinary ineffections
* vaginal prolabs
* qronical lung disease
* psychiatric diseases
* other neurological diseases
* do not speak Danish

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-01; Study Completion 2001-09

PRIMARY OUTCOMES:
Quality of Life parameters (SF-36, IIQ)

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid G Tibaek, MSc., Pt, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Copenhagen University Hospital, Glostrup, Glostrup Municipality, Denmark

REFERENCES:
- [Result] Tibaek S, Jensen R, Lindskov G, Jensen M. Can quality of life be improved by pelvic floor muscle training in women with urinary incontinence after ischemic stroke? A randomised, controlled and blinded study. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):117-23; discussion 123. doi: 10.1007/s00192-004-1124-1. Epub 2004 Jan 31. PMID 15014939
- [Result] Tibaek S, Gard G, Jensen R. Pelvic floor muscle training is effective in women with urinary incontinence after stroke: a randomised, controlled and blinded study. Neurourol Urodyn. 2005;24(4):348-57. doi: 10.1002/nau.20134. PMID 15791633
- [Result] Tibaek S, Gard G, Jensen R. Is there a long-lasting effect of pelvic floor muscle training in women with urinary incontinence after ischemic stroke? A 6-month follow-up study. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Mar;18(3):281-7. doi: 10.1007/s00192-006-0137-3. Epub 2006 Jun 28. PMID 16673051